CLINICAL TRIAL: NCT01781286
Title: The Beneficial Effects of Protein-rich, Afternoon Snacks on Appetite Control, Satiety, and Reward-driven Eating Behavior in Young People
Brief Title: The Beneficial Effects of Healthy Snacks on Appetite Control, Satiety, and Reward-driven Eating Behavior in Young People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Collaborators: Solae, LLC (Industry)
Responsible Party: Principal Investigator, Heather Leidy, Tenure-track Assistant Professor, Heather J Leidy, PhD, University of Missouri-Columbia
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 00039414
Record Dates: First submitted 2013-01-09; First posted 2013-01-31 (Estimated); Results first posted 2018-07-23 (Actual); Last update posted 2018-07-23 (Actual); Status verified 2018-07

CONDITIONS: Obesity
Keywords: Obesity; Snacking; Appetite; Protein; Soy; Reward driven eating; Satiety
MeSH Terms: conditions — Obesity | interventions — Diet, Protein-Restricted

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- High Protein (Active Comparator): Higher Protein Soy-based Snacks
  Interventions: Behavioral: High Protein
- Low Protein (Active Comparator): Typical, Low Protein Snacks
  Interventions: Behavioral: Low Protein
- No Snack (No Intervention): No Snack

INTERVENTIONS:
Behavioral: High Protein — 250 kcal; 40% Protein; 40% Carbohydrate; 20% Fat
  Arms: High Protein
Behavioral: Low Protein — 5% Protein; 50% Carbohydrates; 45% Fat
  Arms: Low Protein

SUMMARY:
The purpose of this study is to examine the effects of normal vs. protein-rich afternoon snacks on appetite control, satiety, and reward-driven eating (particularly in the evening) in young people. Indices of attention and mood will also be assessed.

Study hypotheses include the following:

1. The consumption of a high-protein, soy-rich afternoon snack will lead to significant improvements in appetite control and satiety, reductions in food motivation and reward, and will delay the drive to eat in normal to overweight young people.
2. The consumption of a high-protein, soy-rich afternoon snack will lead to reduced unhealthy, evening snacking, particularly on foods high in fat and/or sugar, in normal to overweight young people.
3. The daily consumption of a high-protein, soy-rich afternoon snack will lead to significant improvements in afternoon alertness, concentration, fatigue, and well-being in normal to overweight young people.

DETAILED DESCRIPTION:
Forty adolescents will participate in the following randomized crossover-design study. Prior to the start of the study, the participants will be asked to document their habitual breakfast, lunch, and afternoon snack times. The snack patterns and associated testing days will be scheduled so that each participant consumes the afternoon snack (or refrains from snacking) 3 hours after lunch; however, the time of day when this occurs is based on the participant's previous, habitual snack time. Once this is determined, each participant will randomly acclimate to the following snack pattern for 3 consecutive days: 1) Higher Protein Soy-based Snacks (250 kcal; 40% Protein; 40% Carbohydrates; 20% Fat); 2) Typical, Low Protein Snacks (5% Protein; 50% Carbohydrates; 45% Fat); and 3) No Snack.

On day 4, the participants will consume a standard breakfast, at home, and lunch, at school, and will come in to our facility 1 hour prior to their habitual snack time. The participants will be placed in a window-less, comfortable room, void of all time cues. They will be informed that they will remain in this room for the next 6 hours. The participants will begin the testing day by completing baseline questionnaires assessing appetite, satiety, mood, and cognitive function. A brain scan will be completed using functional magnetic resonance imaging (fMRI) to identify brain activation patterns in response to food stimuli. Following the fMRI scan, the respective snack will be given to the participants; they will have 15 minutes to eat the snack. A second fMRI scan will then be performed. The participants will continue to complete the previous questionnaires until they voluntarily choose to eat. At this time, the volunteers will be presented with an 'all you can eat' snack buffet. They will be permitted to eat as much or as little as they would like to eat over the next 3-hour period. The participants will remain in the facility until the full 8-hour testing day is completed, regardless of when they requested to eat. Following the 6 hours, the participants will be permitted to leave the facility.

ELIGIBILITY:
Inclusion Criteria:

* Age range 13-19 years
* Normal to overweight (BMI: 50-85th percentile for BMI for age or BMI: 18-29.9 kg/m2)
* No metabolic, psychological, or neurological diseases/conditions
* Not currently or previously on a weight loss or other special diet (in the past 6 months)
* Not clinically diagnosed with an eating disorder
* Habitually eat (i.e., at least 5 times/week) breakfast between 7:00-9:00 am, lunch between 11:00 am-1:00 pm, an afternoon snack between 2:00-4:00 pm, and dinner
* No food allergies or intolerances to soy products
* Rates the overall liking of the study snack foods higher than "Neither Like nor Dislike" on the screening palatability questionnaire
* Right handed

Exclusion Criteria:

* Age 12 years or younger, or 20 years or older
* Underweight or Obese (below 50th or above 85th percentile for BMI for age, or BMI below 18 or above 29.9 kg/m2)
* Any metabolic, psychological, or neurological diseases/conditions
* Currently or previously on a weight loss or other special diet (in the past 6 months)
* Clinically diagnosed with an eating disorder
* Does not habitually eat (i.e., at least 5 times/week) breakfast between 7:00-9:00 am, lunch between 11:00 am-1:00 pm, an afternoon snack between 2:00-4:00 pm, and dinner
* Food allergies or intolerances to soy products
* Does not rate the overall liking of the study snack foods higher than "Neither Like nor Dislike" on the screening palatability questionnaire
* Not right handed

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 37 (Actual)
Dates: Start 2013-01; Primary Completion 2013-10 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heather J Leidy, PhD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri-Columbia, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Leidy HJ, Todd CB, Zino AZ, Immel JE, Mukherjea R, Shafer RS, Ortinau LC, Braun M. Consuming High-Protein Soy Snacks Affects Appetite Control, Satiety, and Diet Quality in Young People and Influences Select Aspects of Mood and Cognition. J Nutr. 2015 Jul;145(7):1614-22. doi: 10.3945/jn.115.212092. Epub 2015 May 20. PMID 25995282

RESULTS

PARTICIPANT FLOW:
Groups:
- High Fat Snack > No Snack > High Protein Snack: 8 Participants began testing procedures but only 31 completed all procedures. Each participant was randomly acclimated to the following snack patterns for 3 consecutive days: 1) Typical, Low Protein Snacks (5% Protein; 50% Carbohydrates; 45% Fat); 2) No Snack and 3) Higher Protein Soy-based Snacks (250 kcal; 40% Protein; 40% Carbohydrates; 20% Fat). On day 4, participants completed all testing day procedures outlined in the study description. Three participants signed the consent form but never began testing procedures. One dropped out before completing the second testing day and another before the third. Upon completion of all thirty two participants, one was later found to be noncompliant with testing day procedures.
- High Fat Snack > High Protein Snack > No Snack: 4 Participants began testing procedures but only 31 completed all procedures. Each participant was randomly acclimated to the following snack patterns for 3 consecutive days: 1) Typical, Low Protein Snacks (5% Protein; 50% Carbohydrates; 45% Fat); 2) Higher Protein Soy-based Snacks (250 kcal; 40% Protein; 40% Carbohydrates; 20% Fat) and 3) No Snack. On day 4, participants completed all testing day procedures outlined in the study description. Three participants signed the consent form but never began testing procedures. One dropped out before completing the second testing day and another before the third. Upon completion of all thirty two participants, one was later found to be noncompliant with testing day procedures.
- No Snack > High Protein Snack > High Fat Snack: 9 Participants began testing procedures but only 31 completed all procedures. Each participant was randomly acclimated to the following snack patterns for 3 consecutive days: 1) No Snack; 2) Higher Protein Soy-based Snacks (250 kcal; 40% Protein; 40% Carbohydrates; 20% Fat) and 3) Typical, Low Protein Snacks (5% Protein; 50% Carbohydrates; 45% Fat). On day 4, participants completed all testing day procedures outlined in the study description. Three participants signed the consent form but never began testing procedures. One dropped out before completing the second testing day and another before the third. Upon completion of all thirty two participants, one was later found to be noncompliant with testing day procedures.
- No Snack > High Fat Snack > High Protein Snack: 8 Participants began testing procedures but only 31 completed all procedures. Each participant was randomly acclimated to the following snack patterns for 3 consecutive days: 1) No Snack; 2) Typical, Low Protein Snacks (5% Protein; 50% Carbohydrates; 45% Fat and 3) Higher Protein Soy-based Snacks (250 kcal; 40% Protein; 40% Carbohydrates; 20% Fat). On day 4, participants completed all testing day procedures outlined in the study description. Three participants signed the consent form but never began testing procedures. One dropped out before completing the second testing day and another before the third. Upon completion of all thirty two participants, one was later found to be noncompliant with testing day procedures.
- High Protein Snack > No Snack > High Fat Snack: 6 Participants began testing procedures but only 31 completed all procedures. Each participant was randomly acclimated to the following snack patterns for 3 consecutive days: 1) Higher Protein Soy-based Snacks (250 kcal; 40% Protein; 40% Carbohydrates; 20% Fat); 2) No Snack and 3) Typical, Low Protein Snacks (5% Protein; 50% Carbohydrates; 45% Fat. On day 4, participants completed all testing day procedures outlined in the study description. Three participants signed the consent form but never began testing procedures. One dropped out before completing the second testing day and another before the third. Upon completion of all thirty two participants, one was later found to be noncompliant with testing day procedures.
- High Protein Snack > High Fat Snack > No Snack: 3 Participants began testing procedures but only 31 completed all procedures. Each participant was randomly acclimated to the following snack patterns for 3 consecutive days: 1) Higher Protein Soy-based Snacks (250 kcal; 40% Protein; 40% Carbohydrates; 20% Fat); 2) Typical, Low Protein Snacks (5% Protein; 50% Carbohydrates; 45% Fat and 3) No Snack. On day 4, participants completed all testing day procedures outlined in the study description. Three participants signed the consent form but never began testing procedures. One dropped out before completing the second testing day and another before the third. Upon completion of all thirty two participants, one was later found to be noncompliant with testing day procedures.
Period: Overall Study
Arm/Group | High Fat Snack > No Snack > High Protein Snack | High Fat Snack > High Protein Snack > No Snack | No Snack > High Protein Snack > High Fat Snack | No Snack > High Fat Snack > High Protein Snack | High Protein Snack > No Snack > High Fat Snack | High Protein Snack > High Fat Snack > No Snack
Started | 7 | 4 | 9 | 8 | 6 | 3
Started 1st Intervention | 6 | 4 | 9 | 8 | 6 | 2
Started 2nd Intervention | 5 | 4 | 9 | 8 | 6 | 2
Started 3rd Intervention | 5 | 4 | 7 | 7 | 6 | 2
Completed | 5 | 4 | 7 | 7 | 6 | 2
Not Completed | 2 | 0 | 2 | 1 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Time Constraints | 2 | 0 | 2 | 0 | 0 | 0
Not completed — Noncompliance | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Each participant was randomly acclimated to the following snack patterns for 3 consecutive days: 1) Higher Protein Soy-based Snacks (250 kcal; 40% Protein; 40% Carbohydrates; 20% Fat); 2) Typical, Low Protein Snacks (5% Protein; 50% Carbohydrates; 45% Fat); and 3) No Snack. On day 4, participants completed all testing day procedures outlined in the study description.
Arm/Group | All Study Participants
Number analyzed (Participants) | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 17 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 15
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 31
Height [Mean (Standard Deviation); unit: centimeters] | 171 (2)
Weight [Mean (Standard Deviation); unit: kilograms] | 65.6 (2.1)
BMI (kg/m2) [Mean (Standard Deviation); unit: kg/m2] | 22.3 (0.4)
BMI (%) [Mean (Standard Deviation); unit: Percentile] | 58.4 (4.4)
Frequency of Snacking [Mean (Standard Deviation); unit: days/week] | 6 (1)
Commonly consumed chips/crackers as a snack [Number; unit: % of total participants] | 64
Commonly consumed fruit as a snack [Number; unit: % of total participants] | 61
Commonly consumed cereal as a snack [Number; unit: % of total participants] | 25

OUTCOME MEASURES:

1. Primary Outcome: Time to Dinner Request
Description: The participants will be asked whether they would like to request a dinner buffet throughout the 5 h post-snack period. When the response is "Yes, I want to eat right now", the time from snack consumption will be recorded.
Time Frame: 1 Day
Measure: Mean (Standard Error); unit: minutes
Groups:
- High Fat (Low Protein): Typical High Fat (Low Protein) Snacks
  5% Protein; 50% Carbohydrates; 45% Fat
- No Snack: No snack was received
Arm/Group | High Protein | High Fat (Low Protein) | No Snack
Number analyzed (Participants) | 31 | 31 | 31
minutes | 158 (7) | 150 (6) | 140 (6)

2. Secondary Outcome: Appetite Questionnaires
Description: Computerized questionnaires, assessing perceived sensations of appetite will be completed throughout the testing days. The questionnaires contain visual analog scales incorporating a 100 mm horizontal line rating scale for each response. The questions are worded as "how strong is your feeling of" with anchors of "not all" (scored as 0 out of 100) to "extremely" (scored as 100 out of 100). The following questions will be incorporated as 1 composite score ((Questions 1 + 3 + 4 - 2)/4) multiplied by the 300 minutes (a max of 30,000 mm*min and a minimum of -30,000 mm*min):
  1. How strong is your feeling of hunger?
  2. How strong is your feeling of being full?
  3. How strong is your desire to eat?
  4. How much food could you consume right now?
  The Adaptive Visual Analog Scale Software (Neurobehavioral Research Laboratory and Clinic; San Antonio, TX) was used for these assessments.
Time Frame: 0 min, + 30 min, +60 min, +90 min, +120 min, +150 min, +180 min, +210 min, +240 min, +270 min, +300 min
Measure: Mean (Standard Error); unit: mm*min
Groups:
- High Fat (Low Protein): Typical, High Fat (Low Protein) Snacks
  5% Protein; 50% Carbohydrates; 45% Fat
Arm/Group | High Protein | High Fat (Low Protein) | No Snack
Number analyzed (Participants) | 31 | 31 | 31
mm*min | -5500 (1000) | -3000 (1000) | 3000 (1000)

3. Secondary Outcome: Snack Palatability and Perception Questionnaires
Description: Computerized questionnaires, assessing snack palatability and perceptions of the snack will be completed during screening and after the first and last bite of each snack during the acclimation and testing days. The questionnaires contain visual analog scales incorporating a 100 mm horizontal line rating scale for each response. The questions are worded as "how strong is your feeling of" with anchors of "not all" (scores 0 out of 100) to "extremely" (scores 100 out of 100). The questions assess snack appearance, smell, flavor, texture (feel), liking.
  The Adaptive Visual Analog Scale Software (Neurobehavioral Research Laboratory and Clinic; San Antonio, TX) was used for these assessments.
Time Frame: 5 min
Measure: Mean (Standard Error); unit: millimeters
Arm/Group | High Protein | High Fat (Low Protein) | No Snack
Number analyzed (Participants) | 31 | 31 | 31
millimeters | 69 (4) | 80 (3) | NA (NA) — No snack was consumed. Therefore, palatability could not be assessed.

4. Secondary Outcome: Attention & Memory Questionnaires
Description: Cognitive function will be assessed immediately before (-30 min) and 60 min post-snack using the lap-top based Cantab® computerized assessment system. This program consisted of a core battery of tests grouped into main categories including 1) Working Memory; 2) Reasoning; 3) Executive Function; 4) Reaction Time; 5) Sustained Attention; 6) Cognitive Flexibility; and 7) Processing Speed. This program has been used in our previous breakfast studies with success. A greater raw score for working memory, reasoning, executive function, sustained attention, and cognitive flexibility is considered to be greater performance. A lower score for reaction time and processing speed is considered to be greater performance. The raw scores are determined by Cantab® computerized assessment system. Therefore, maximum and minimum values for each test are unknown.
Time Frame: 90 min
Measure: Mean (Standard Error); unit: Units on a Scale
Groups:
- No Snack: No snack was received (0 kJ)
Arm/Group | High Protein | High Fat (Low Protein) | No Snack
Number analyzed (Participants) | 31 | 31 | 31
Units on a Scale
  Working Memory (pre-snack) | 102 (3) | 106 (2) | 105 (2)
  Reasoning (pre-snack) | 107 (2) | 108 (2) | 105 (2)
  Executive Function (pre-snack) | 108 (3) | 114 (2) | 112 (2)
  Reaction Time (pre-snack) | 106 (3) | 107 (3) | 103 (2)
  Sustained Attention (pre-snack) | 102 (2) | 105 (1) | 106 (1)
  Cognitive Flexibility (pre-snack) | 108 (4) | 114 (2) | 110 (2)
  Processing Speed (pre-snack) | 110 (3) | 114 (3) | 112 (3)
  Working Memory (post-snack) | 106 (2) | 106 (2) | 104 (2)
  Reasoning (post-snack) | 106 (2) | 110 (2) | 109 (2)
  Executive function (post-snack) | 113 (2) | 116 (2) | 112 (2)
  Reaction Time (post-snack) | 103 (3) | 107 (3) | 105 (3)
  Sustained Attention (post-snack) | 106 (1) | 105 (1) | 104 (2)
  Cognitive Flexibility (post-snack) | 112 (3) | 116 (2) | 112 (2)
  Processing Speed (post-snack) | 118 (3) | 122 (4) | 119 (3)

5. Secondary Outcome: Mood-state Questionnaires
Description: Indices of mood state will be assessed immediately before and 60 min post-snack using the on-line, Profile of Mood States, 2nd Edition (POMS2). This program consisted of a core battery of tests with the following sub-categories 1) Tension; 2) Depression; 3) Anger; 4) Vigor; 5) Fatigue; 6) Confusion; and 7) Friendliness. Outcomes are scored as a T-score which could be a minimum of zero with no upper limit. A lower score represents a more positive mood state and a higher score represents a more negative mood state.
Time Frame: -30 min, +60 min
Measure: Mean (Standard Error); unit: T-Score
Arm/Group | High Protein | High Fat (Low Protein) | No Snack
Number analyzed (Participants) | 31 | 31 | 31
T-Score
  Confusion (-30 min) | 43.5 (0.7) | 42.1 (0.4) | 42.3 (0.6)
  Confusion (+60 min) | 42.2 (0.5) | 41.8 (0.4) | 42.4 (0.5)
  Fatigue (-30 min) | 47.4 (1.4) | 48.2 (1.3) | 49.6 (1.4)
  Fatigue (+60 min) | 47.9 (1.3) | 47.2 (1.2) | 50 (1.2)
  Tension (-30 min | 42.8 (0.5) | 42.4 (0.4) | 43.2 (0.7)
  Tension (+60 min) | 42.2 (0.4) | 42.1 (0.4) | 41.9 (0.3)
  Vigor (-30 min) | 45.6 (1.8) | 44.2 (1.8) | 45.0 (1.2)
  Vigor (+60 min) | 44.2 (1.9) | 43.2 (1.6) | 42.3 (1.5)
  Anger (-30 min) | 41.7 (0.5) | 41.3 (0.4) | 41.5 (0.5)
  Anger (+60 min) | 40.8 (0.3) | 40.5 (0.2) | 41.5 (0.6)
  Depression (-30 min) | 43.5 (0.6) | 42.8 (0.5) | 43.1 (0.6)
  Depression (+60 min) | 55.1 (12.5) | 42.5 (0.2) | 43 (0.5)
  Friendliness (-30 min) | 45.8 (1.6) | 45.3 (1.6) | 46.8 (1.4)
  Friendliness (+60 min) | 44.4 (1.6) | 44.0 (1.7) | 43.3 (1.5)

6. Secondary Outcome: Energy Intake
Description: Post-snack energy intake will be assessed through ad libitum dinner and snacking assessments. The ad libitum dinner will contain approximately 2,000 kcal and will consist of a chicken, rice, and stir-fry meal, chips, chocolate mints, ice tea, and water. The dinner meal will be consumed in the testing facility. The participants will be instructed to eat as much as or as little as they choose over a 30 min period. All contents will be weighed before the dinner and any remains will be re-weighed afterwards to determine the type and quantity of foods consumed.
  The ad libitum evening snacks will contain 3,000 kcal and will include common snack foods. After the testing day is complete, the participants will take the snack packout home and consume any of the foods he/she chooses until going to bed. All contents will be weighed before the packout and any remains will be re-weighed afterwards to determine the type and quantity of foods consumed.
Time Frame: +300 min, 24 h
Measure: Mean (Standard Error); unit: kilojoules
Arm/Group | High Protein | High Fat (Low Protein) | No Snack
Number analyzed (Participants) | 31 | 31 | 31
kilojoules | 3080 (230) | 3370 (290) | 3170 (240)

ADVERSE EVENTS:
Time Frame: 4 months (May 2013 through August 2013).
Arm/Group | High Protein | Low Protein | No Snack
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/31 | 0/31
Other Adverse Events (participants affected / at risk) | 0/31 | 0/31 | 0/31

LIMITATIONS AND CAVEATS:
Menstrual cycle was not controlled for within the female participants. However, menstrual cyclicity varied between testing days and between participants, thus, reducing any systematic bias/effect.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No